CLINICAL TRIAL: NCT00001418
Title: Positron Emission Tomographic (PET) Scanning of Sympathetic Innervation and Function in Patients With Neurocardiologic Disorders
Brief Title: PET Scan in Patients With Neurocardiologic Disorders
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 940186; 94-N-0186
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-08

CONDITIONS: Autonomic Nervous System Diseases
Keywords: Sympathetic Nervous System; Dysautonomias; Postural Tachycardia Syndrome; Neurocardiogenic Syncope; Hypernoradrenergic Hypertension; Sympathectomy; Fluorodopamine; Positron Emission Tomography; Norepinephrine; Dopamine; Neurocardiologic Disorder
MeSH Terms: conditions — Autonomic Nervous System Diseases; Postural Orthostatic Tachycardia Syndrome; Syncope, Vasovagal

SUMMARY:
This study is designed to use PET scans in order to measure activity of the sympathetic nervous system. The sympathetic nervous system is the portion of the nervous system that maintains a normal supply of blood and fuel to organs during stressful situations.

PET scan or Positron Emission Tomography is an advanced form of an X-ray. It is used to detect radioactive substances in the body. During this study researchers plan to inject small amounts of the radioactive drug fluorodopamine into patients. Fluorodopamine is very similar to the chemicals found in the sympathetic nervous system. It can attach to sympathetic nerve endings and allow researchers to view them with the aid of a PET scan. One area of the body with many sympathetic nerve endings is the heart. After giving a dose of fluorodopamine, researchers will be able to visualize all of the sympathetic nerve endings involved in the activity of the heart. In addition, this diagnostic test will help researchers detect abnormalities of the nervous system of patient's hearts.

DETAILED DESCRIPTION:
This project applies positron emission tomographic (PET) scanning after administration of 6-[18F]fluorodopamine ([18F]-6F-DA) to visualize sympathetic innervation and function in patients with neurocardiologic disorders. Patients undergo infusion of [18F]-6F-DA, followed by PET scanning of one or more body regions. Patients may also undergo PET scanning after administration of [13N]-ammonia, to assess regional perfusion; regional blood sampling (including sampling from the coronary sinus or great cardiac vein) during infusion of [3H]-l-norepinephrine ([3H]-NE), to assess the kinetics and metabolism of NE; or magnetic resonance imaging (MRI) to delineate the ventricular myocardium. PET scanning after [18F]-6F-DA administration, in conjunction with other clinical assessment tools, should provide comprehensive information about regional sympathoneural innervation and function in neurocardiologic disorders.

ELIGIBILITY:
INCLUSION CRITERIA:

The subjects are adult patients in one of the following diagnostic categories: coronary heart disease or chest pain and normal coronary arteries; myocardial dysfunction or failure; hypertension; or dysautonomia. Groups of appropriately matched healthy volunteers are studied concurrently as controls.

EXCLUSION CRITERIA:

Minors are excluded.

Subjects in whom anatomic factors complicate vascular access are excluded.

Subjects who are not expected clinically to tolerate recumbency during the procedures are excluded.

Pregnant or lactating women are excluded.

Cardiology patients may be tested while off their usual medications. In this situation, the patients will be inpatients on the cardiology ward, managed clinically by staff of the Cardiology Branch, DIR, NHLBI. Hypertensives will be tested afer having discontinued anti-hypertensive medications for up to two weeks.

Patients who must take medications continually in the following categories are excluded: anticoagulants, tricyclic antidepressants, barbiturates, aspirin, acetaminophen.

Patients unable to discontinue nicotine or alcohol temporarily are excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 335
Dates: Start 1994-07; Study Completion 2004-08

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States